CLINICAL TRIAL: NCT06754709
Title: Evaluation of the Levels of O-GlcNAcylation of Cardiac and Blood Proteins in Paediatric Cardiac Surgery and Identification of Therapeutic Targets
Brief Title: Evaluation of Blood and Cardiac Protein O-GlcNAcylation Levels in Cardiac Surgery in Children
Acronym: CardiOGlcNAc
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC24_0572
Record Dates: First submitted 2024-12-23; First posted 2025-01-01 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Cardiac Surgery; Extracorporeal Circulation; Complications; Metabolism; Low Cardiac Output
Keywords: cardiac surgery; extracorporeal circulation; metabolism; low cardiac output; O-GlcNAcylation,; systemic inflammatory response syndrome
MeSH Terms: conditions — Cardiac Output, Low; Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample, cardiac tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac surgery with extracorporeal circulation: Children aged between 0 and 17 undergoing cardiac surgery with extracorporeal circulation.
  The children will have blood samples taken at the same time as the samples already taken for all the children as part of the intra- and post-operative management of cardiac surgery. If necessary, the resection of cardiac tissue planned for cardiac surgery will be preserved for the study. Patients' administrative data will be collected at the time of sampling and anonymised. Medical data will be collected retrospectively from the medical record. Patients will be monitored as part of the post-operative cardiac surgery network and data will be collected retrospectively from the patient's file.
  Western blot analysis (measurement of O-GlcNAcylation) will be carried out as soon as a sufficient number of samples are available in the bio-collection (generally by 15 samples)

SUMMARY:
Cardiac surgery requires the use of extracorporeal circulation (ECC). Age-related differences in inflammatory response, the greater susceptibility of immature organ systems to injury and the larger ratio of extracorporeal circuitry to patient size make younger and smaller patients more vulnerable to organ injury. The main problem associated with ECC in neonates and infants is the duration of ECC due to heavier surgeries leading to a prolonged inflammatory state resulting in capillary leak syndrome, low cardiac output syndrome and organ dysfunction, resulting in higher morbidity and mortality. The means of limiting this inflammatory response remain limited. Future studies should aim to address new post-ECC prophylactic targets to improve myocardial and endothelial function. Cardiac metabolism is an important area of research because it plays a central role in maintaining cardiac function under stress. The study of O-GlcNAcylation could therefore be an interesting therapeutic target, given the beneficial role of its stimulation in acute stress situations, as demonstrated in sepsis.

DETAILED DESCRIPTION:
Extracorporeal circulation (ECC) is a circuit that provides circulatory assistance to facilitate surgical access to a bloodless and, in some cases (in the case of cardioplegia) immobile operating field. This strategy has led to technical and procedural advances in cardiothoracic surgery that would have been unthinkable without bypass surgery. ECC leads to systemic inflammatory response syndrome and is associated with postoperative complications, including myocardial dysfunction, respiratory failure, acute renal failure, neurological dysfunction, coagulation disorders and, finally, multivisceral failure. Numerous data suggest that inflammation and oxidative stress occur shortly after the start of bypass surgery and progress over time. ECC-induced SIRS, similar to sepsis, leads to stimulation and activation of endothelial cells. Circulating pro-inflammatory cytokines can also directly stimulate endothelial cells, resulting in a pathological increase in permeability leading to the development of capillary leak syndrome, causing tissue oedema and impaired oxygen utilisation leading to multiple organ dysfunctions. Clinical practice has shown that the majority of infants suffer haemodynamic failure within 4 to 8 hours of the operation. This failure could be related to a state of vasodilatation (capillary leakage) and/or a low cardiac output syndrome. The timing of the onset of this failure correlates with peak cytokine secretion. The risk factors for severe SIRS in paediatric cardiac surgery are low weight, heart disease with an intra-cardiac right-left shunt, the duration of aortic clamping and the length of the bypass operation. This state of vasoplegia is associated with an increase in lactate production, reflecting an imbalance between organ oxygen demand and supply, an increase in amine requirements and an increase in invasive ventilation time. In many cases, vasoplegia is associated with low cardiac output syndrome. This syndrome is the most common post-operative complication in paediatric cardiac surgery. Twenty-five to sixty per cent of newborns develop low cardiac output syndrome (LCOS) in the 6 to 18 hours following surgery, with mortality occurring in 20% of cases. Current means of limiting post-CEC SIRS remain limited. The understanding of inflammatory processes and the interaction between humoral factors and the cellular immune response has progressed rapidly over the last decade. Multiple anti-inflammatory strategies have been applied in the past, significantly reducing cytokine levels without improving clinical outcome. This means that the amplitude of inflammatory cytokine secretion does not directly predict patient outcome. Future studies should aim to address new post-CEC prophylactic targets to improve myocardial and endothelial function. Cardiac metabolism is an important area of research because it plays a central role in maintaining cardiac function under stress. In recent years, there has been considerable interest in O-GlcNAcylation, a post-translational modification of proteins, as it plays a key role in regulating cellular metabolism and the ability to adapt to stress and cell survival. O-N-acetyl glucosaminylation, more simply known as O-GlcNAcylation, is a ubiquitous, rapid and reversible post-translational modification involving the addition of a monosaccharide: ß-D-N-acetylglucosamine to the serine and threonine residues of proteins. In physiological conditions, some of the glucose entering the cell is directed towards the hexosamine biosynthesis pathway (VBH), which leads to the production of UDP-GlcNAc, used by O-GlcNAc transferase (OGT) to O-GlcNAcylate proteins. The reverse reaction is catalysed by O-GlcNAcase (OGA). VBH is at the crossroads of several cellular metabolic pathways (glucose, acetyl-CoA, glutamine, uridine and ATP) and O-GlcNAcylation is considered to be a metabolic sensor. The number of O-GlcNAcylated targets (+3000 proteins) bears witness to the involvement of this modification in various cellular functions. O-GlcNAc levels are finely modulated according to the cell's metabolic environment, enabling it to adapt to stress. This last point is particularly important as metabolism changes during development and during CEC, which impacts the hexosamine biosynthesis pathway and therefore O-GlcNAcylation. O-GlcNAcylation is particularly difficult to study at cardiac level, but the investigators have shown that there is a close correlation between blood (whole blood) and cardiac O-GlcNAc levels in rats. Preliminary data in rats have shown that O-GlcNAcylation levels decrease during bypass surgery and that there is an interest in increasing O-GlcNAcylation levels during bypass surgery in order to reduce organ failure, but no human data have been published in this context.

ELIGIBILITY:
Inclusion Criteria:

* Age from 0 to 17 years at the time of sampling
* Children undergoing CEC for cardiac surgery
* Signed bio-collection consent

Exclusion Criteria:

* Children with an infection
* Children with fever
* Children with an immune deficiency
* Children with autoimmune disease
* Children with metabolic disease
* Children with haematological diseases
* Children with a genetic disease
* Unsigned consent
* Refusal by parents or child

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged between 0 and 17 undergoing cardiac surgery with extracorporeal circulation
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2034-01-31 (Estimated); Study Completion 2035-01-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of O-GlcNAcylation levels in cardiac surgery in children | From start of the surgery to 12 hours after start of the surgery
  To evaluate the evolution of O-GlcNAcylation levels in pre-per-post extracorporeal circulation in children

SECONDARY OUTCOMES:
Analysis of a potential link between O-GlcNAcylation levels and the prognosis of patients after cardiac surgery | Up to 6 years after inclusion
  To study the correlation between blood and cardiac O-GlcNAcylation levels and patient prognosis

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: Undecided